CLINICAL TRIAL: NCT04761185
Title: Phase I Clinical Human Tolerability Test of Raltitrexed in Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Raltitrexed in HIPEC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, MD, PHD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-RAL
Record Dates: First submitted 2021-01-05; First posted 2021-02-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Raltitrexed; HIPEC
Keywords: Colorectal Cancer; Raltitrexed; HIPEC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — raltitrexed; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: Employing a standard 3+3 dose-escalation design, RTX was administered at doses ranging from 3 to 9 mg/m2 during HIPEC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIPEC using Raltitrexed (Experimental)
  Interventions: Drug: Raltitrexed

INTERVENTIONS:
Drug: Raltitrexed — The RTX-HIPEC protocol used a modified Fibonacci dose escalation method with 7 dose levels (3, 4, 5, 6, 7, 8, 9 mg/m2)
  Other Names: HIPEC

SUMMARY:
To evaluate the tolerance of patients with colorectal cancer to hyperthermic intraperitoneal chemotherapy with Raltitrexed, to determine the dose limiting toxicity and maximum tolerated dose.

DETAILED DESCRIPTION:
All patients with CRC-PM who underwent CRS at the Department of Colorectal Surgery, Fudan University Shanghai Cancer Center between September 2020 and November 2024 were enrolled as part of the classical 3+3 dose-escalation phase I trial, and within a later expansion cohort. Initially, 3 patients were sequentially evaluated for DLTs at each dose level. The MTD was defined as the highest dose in cohorts where ≦1 patients experienced DLT. Thereafter, additional patients were enrolled in an expansion cohort to determined RP2D. The recommended phase II dose (RP2D) was the highest dose level which no patients had a DLT. The RTX-HIPEC protocol used a modified Fibonacci dose escalation method with 7 dose levels (3, 4, 5, 6, 7, 8, 9 mg/m2).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75 (including 18 and 75), regardless of gender;
2. ECOG score ≤1;
3. Patients with colorectal adenocarcinoma/mucinous adenocarcinoma/signet ring cell carcinoma/mucinous tumor confirmed by histopathology;
4. The laboratory test results within 1 week before treatment meet the following conditions:

   White blood cell (WBC) ≥ 4.0×109 /L;Neutrophil count (ANC) ≥ 1.8×109 /L;Platelet (PLT) ≥ 100×109/L;Hemoglobin (Hb) ≥ 80 g/L;Serum total bilirubin (TB) ≤ 1.5×ULN;Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT)≤ 2.5×ULN;Blood urea nitrogen (BUN) and blood creatinine (Cr) ≤ 1.5×ULN;
5. Patients voluntarily participate in this study, sign written informed consent, have good compliance and are willing to cooperate with the follow-up.

Exclusion Criteria:

1. Patients with severe complications were considered to be intolerant of postoperative chemotherapy;
2. Previous or concurrent malignancy, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin;
3. Patients with peptic ulcer, gastrointestinal dynamic obstruction, severe active bleeding of the digestive tract, and perforation of the digestive tract;
4. Those with a history of allergy to the drug components or metabolites in the program;
5. A history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
6. had any heart disease, including :(1) angina;(2) Arrhythmia requiring medical treatment or clinically significant;(3) Myocardial infarction;(4) Heart failure;(5) any other heart disease deemed unfit to participate in this study by the researcher;
7. Female patients during pregnancy and lactation, female patients with fertility and positive test of baseline pregnancy or female patients of childbearing age who are unwilling to take effective contraceptive measures during the whole test period;
8. The accompanying diseases (including but not limited to hypertension, severe diabetes, active infection, thyroid disease, etc.) that, according to the judgment of the researcher, seriously endanger the safety of the patient or affect the completion of the study;
9. A past history of neurological or mental disorders, such as major depression, epilepsy, or dementia, that clearly affect study disclosure or follow-up evaluation;
10. Participate in other clinical trials within 30 days of enrollment and receive research drugs and any concomitant treatment containing research drugs;
11. Other conditions in which the investigator considers it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose limiting toxicity. | Within 21 days post-treatment
  to determine dose-limiting toxicity
tolerable dose | Up to 21 days post-treatment
  to determine maximum tolerable dose

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 48 hours after administration
Time to maximum concentration (Tmax) | Up to 48 hours after administration
Area under the drug concentration-time curve from time 0 to the last measurable concentration time point (AUC0-t) | Up to 48 hours after administration
Recurrence-free survival (RFS) | Up to 2 years
  Time from RTX-HIPEC date until progression per RECIST v1.1 as assessed by the investigator at local site, or death due to any cause.
Apparent volume of distribution (Vz/F) and clearance (CLz/F) | Up to 48 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China